CLINICAL TRIAL: NCT06404047
Title: RECOVER-ENERGIZE: A Platform Protocol for Evaluation of Interventions for Exercise Intolerance in Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Brief Title: RECOVER-ENERGIZE Platform Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00112409; OT2HL156812 (NIH); NHLBI Grant to RTI (Other Grant/Funding Number: RTI subcontracting with DCRI)
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Long COVID; Long Covid19; Long Covid-19
Keywords: PASC; Exercise; PEM (post exertional malaise)
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This platform protocol is designed to allocate participants into an appropriate intervention appendix based on their symptoms of exercise intolerance or post-exertional malaise (PEM). Once assigned to an appendix, eligible participants are randomized in a 1:1 ratio to either the study intervention group or a control group.
Who Masked: Outcomes Assessor
Masking Description: Appendix A: Single (Outcomes Assessor masked) The assessor of the primary outcome, Endurance Shuttle Walk Test (ESWT), is blinded.
  Appendix B: None (open label / no masking)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Appendix A - Cardiopulmonary Rehabilitation (Exercise Intolerance) (Experimental): Appendix A is a randomized controlled trial designed to evaluate the effect of a 12-week personalized cardiopulmonary rehabilitation intervention on exercise tolerance in participants with PASC.
  Participants who meet eligibility criteria for Appendix A will be assigned to either Personalized Cardiopulmonary Rehabilitation (study intervention group) or Education (control group) in a 1:1 ratio. The intervention duration is 12 weeks with a follow-up period of 3 months (total study duration of 6 months).
  Anticipated enrollment is 360 participants. Details about Appendix A: Cardiopulmonary Rehabilitation (Exercise Intolerance) are available under NCT06404060.
  Interventions: Behavioral: Personalized Cardiopulmonary Rehabilitation; Other: Education
- Experimental: Appendix B - Structured Pacing (PEM) (Experimental): Appendix B is a randomized controlled trial designed to evaluate the effect of a 12-week Structured Pacing intervention on reducing the symptoms of post-exertional malaise (PEM) in participants with PASC.
  Participants who meet eligibility criteria for Appendix B will be assigned to either Structured Pacing (study intervention group) or Usual Care (control group) in a 1:1 ratio. The intervention duration is 12 weeks with a follow-up period of 3 months (total study duration of 6 months).
  Anticipated enrollment is 300 participants. Details about Appendix B: Structured Pacing (PEM) are available under NCT06404073.
  Interventions: Behavioral: Structured Pacing; Other: Usual Care

INTERVENTIONS:
Behavioral: Personalized Cardiopulmonary Rehabilitation — Participants in this group will complete 2-3 cardiopulmonary rehabilitation sessions per week, for 12 weeks, as tolerated. Rehabilitation sessions are provided by respiratory therapists, exercise physiologists, physical therapists, nurses, or others who have experience and training in either pulmonary or cardiac rehabilitation.
  Rehabilitation sessions (adjusted based on the participant's baseline assessment, symptoms, and progress) last about 1 hour and include education, aerobic exercise, strength, and flexibility training.
  Arms: Experimental: Appendix A - Cardiopulmonary Rehabilitation (Exercise Intolerance)
Behavioral: Structured Pacing — Participants in this group will complete weekly pacing sessions for 12 weeks. Pacing sessions will last about 30 minutes, as tolerated. Each participant will meet with a provider 'pacing coach' who has received study-specific education about PEM and how to create and manage pacing strategies for participants. Sessions include PEM symptom and trigger assessment; task, function and activity analysis; adaptations and modifications.
  Arms: Experimental: Appendix B - Structured Pacing (PEM)
Other: Education — Participants in this group will receive two general education sessions at the start of the intervention with weekly phone/virtual follow-ups from site study staff.
  Arms: Experimental: Appendix A - Cardiopulmonary Rehabilitation (Exercise Intolerance)
Other: Usual Care — Participants in this group will receive basic education about PEM with a weekly call by site study staff for support and communication.
  Arms: Experimental: Appendix B - Structured Pacing (PEM)

SUMMARY:
This is a platform protocol designed to be flexible so that it is suitable for a range of interventions and settings within diverse health care systems and community settings with incorporation into clinical COVID-19 management programs and treatment plans if results achieve key study outcomes.

This protocol is a prospective, multi-center, multi-arm, randomized, controlled platform trial evaluating interventions to address and improve exercise intolerance and post-exertional malaise (PEM) as manifestations of Post-Acute Sequelae of SARS-CoV-2 Infection (PASC).

The focus of this protocol is to assess interventions that can improve exercise capacity, daily activities tolerance, and quality of life in patients with PASC.

DETAILED DESCRIPTION:
Study interventions will be added to the platform protocol as appendices. Each appendix will leverage all elements of the platform protocol, with additional elements described in the individual appendix. Study intervention appendices may be added or removed according to adaptive design and/or emerging evidence.

The platform protocol enrolls participants who meet study eligibility criteria. After completing initial screening assessments, eligible participants are assigned to one of the study intervention appendices that are actively enrolling. Participants must meet certain criteria within a specific appendix in order to be included in that appendix. Once assigned to an appendix, eligible participants are randomized to either the study intervention group or a control group.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of enrollment
2. Previous suspected, probable, or confirmed SARS-CoV-2 infection, as defined by the Pan American Health Organization*

   * Suspected* or probable SARS-CoV-2 infection will only be allowed if it occurred before May 1, 2021, and will be limited to no more than 10% of the study population. Otherwise, confirmed cases are required.

   Suspected case of SARS-CoV-2 infection - Three options, A through C:

   A. A person who meets the clinical OR epidemiological criteria. Clinical criteria: Acute onset of fever AND cough (influenza-like illness) OR Acute onset of ANY THREE OR MORE of the following signs or symptoms: fever, cough, general, weakness/fatigue, headache, myalgia, sore throat, coryza, dyspnea, nausea, diarrhea, anorexia. Epidemiological criteria: Contact of a probable or confirmed case or linked to a COVID-19 cluster; or B. Acute respiratory infection with history of fever or measured fever of ≥ 38°C; and cough; with onset within the last 10 days; and who requires hospitalization; or C. With no clinical signs or symptoms, NOR meeting epidemiologic criteria with a positive professional use or self-test SARS-CoV-2 Antigen-Rapid Diagnostic Test.

   Probable case of SARS-CoV-2 infection:

   A. A patient who meets clinical criteria above AND is a contact of a probable or confirmed case or is linked to a COVID-19 cluster.

   Confirmed case of SARS-CoV-2 infection - Two options, A and B:

   A. A person with a positive nucleic acid amplification test, regardless of clinical criteria OR epidemiological criteria; or B. Meeting clinical criteria AND/OR epidemiological criteria (See suspected case A above for criteria). With a positive professional use or self-test SARS- CoV-2 Antigen-Rapid Diagnostic Test.
3. Self-reported limitation to physical activity due to the presence of symptoms such as fatigue, shortness of breath, and/or PEM following a SARS-CoV-2 infection, that has persisted for at least 12 weeks and is present at the time of consent.
4. Willing, able, and agree to provide informed consent, complete questionnaires and outcome assessments, and participate in the study, including assigned intervention or control and study visits whether remote, hybrid, or in-person.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Known active acute SARS-CoV-2 infection ≤ 4 weeks prior to the consent.
2. Known prior diagnosis of Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS), not related to SARS-CoV-2 infection.
3. Current or recent use (within the last 14 days) of a formal program utilizing one or more of the current study intervention(s) or similar intervention(s) to treat the underlying condition, unless a washout period is permitted per Appendices.
4. Participation in another interventional clinical trial.
5. Any condition that would make the participant, in the opinion of the investigator, unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Total number of participants enrolled in each Appendix | 6 months
  Total number of participants enrolled in each Appendix will be reported. Appendix-specific outcome measure data will be reported under the associated NCT#

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Felker, MD, Study Chair — Duke Clinical Research Institute; Barry Make, MD, Study Chair — National Jewish Health; Lucinda Bateman, MD, Study Chair — Bateman Horne Center; Janna Friedly, MD, MPH, Study Chair — University of Washington
Locations (42):
- United States (42):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Banner University Medical Center Tucson, Tucson, Arizona
  - Stanford University, Stanford, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Yale - New Haven Hospital, New Haven, Connecticut
  - University of Florida College of Medicine Jacksonville, Jacksonville, Florida
  - Innovation Clinical Trials Inc., Miami, Florida
  - Valencia Medical and Research Center, Miami, Florida
  - Grady Memorial Hospital (Emory), Atlanta, Georgia
  - Emory Hope Clinic, Decatur, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - North Shore University HealthSystem/Evanston Hospital, Evanston, Illinois
  - Saint Francis Medical Center, Peoria, Illinois
  - Cedar Valley Clinical Research, Waterloo, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Maine Health Institute of Research, Scarborough, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - NYU Langone Health/Brooklyn Hospital, Brooklyn, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Avera McKennan Hospital & University Health Center, Sioux Falls, South Dakota
  - Southwest Family Medicine Associates, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Vermont Lung Center, University of Vermont, Colchester, Vermont
  - University Physicians and Surgeons, Inc dba Marshall Health, Huntington, West Virginia
  - West Virginia Clinical and Translational Science Institute, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No
The summary of the results will be shared on the study website: https://recovercovid.org/

REFERENCES:
- See also: Related Info — http://recovercovid.org/

DOCUMENTS (1):
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT06404047/ICF_000.pdf